CLINICAL TRIAL: NCT02519075
Title: Diagnostic and Prognostic Role of 11C-Choline PET/CT and DWI MRI for Response Assessment in Patients Affected by Hepatocellular Carcinoma (HCC) and Candidate to TARE
Brief Title: 11C-Choline PET/CT and DWI MRI for Response Assessment of HCC Candidate to TARE
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1386
Record Dates: First submitted 2015-06-26; First posted 2015-08-10 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Hepatocarcinoma
Keywords: Hepatocarcinoma; TARE; response assessment
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — Biopsy specimen
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — Observational study

SUMMARY:
Prospective exploratory study specifically investigating the diagnostic and predictive role of 11C-Choline PET/CT and DWI MRI for response assessment in patients affected by HCC and candidate to TARE. A minimum number of 20 patients will be considered for the analysis.

DETAILED DESCRIPTION:
For the study, all patients with a histological diagnosis of HCC and eligible for TARE, i.e. with liver predominant disease who are not eligible for curative surgery, after multidisciplinary discussion will be included. In all cases, patients will undergo 11C-Choline PET/CT and DWI MRI before starting radioembolization and will be subsequently restaged 3 months after treatment completion. A minimum number of 20 patients will be considered for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients with a histological diagnosis of HCC and eligible for TARE, i.e. with liver predominant disease who are not eligible for curative surgery, after multidisciplinary discussion will be included;
* obtained informed consent

Exclusion Criteria:

* patients age <18 years
* pregnancy or breast-feeding;
* patients affected by other malignancies within the last 3 years;
* disseminated extrahepatic disease;
* severely abnormal excretory liver function tests or ascites suggestive of liver failure;
* hepatopulmonary shunt >20%;
* vascular variants and abnormalities as demonstrated on pre-treatment angiography, which cannot be corrected by embolisation and which lead to reflux of hepatic arterial blood to the stomach, pancreas or bowel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients affected by HCC and referred to our Institution for TARE will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Variation of SUVmax (Maximal Standardized Uptake Value) in patients undergoing TARE for HCC | Change from Baseline in SUVmax up to 3 months after TARE

CONTACTS AND LOCATIONS:
Overall Officials: Egesta Lopci, MD, Principal Investigator — Humanitas Clinical and Research Hospital
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

REFERENCES:
- [Background] Lopci E, Torzilli G, Poretti D, de Neto LJ, Donadon M, Rimassa L, Lanza E, Sabongi JG, Ceriani R, Personeni N, Palmisano A, Pedicini V, Comito T, Scorsetti M, Chiti A. Diagnostic accuracy of (1)(1)C-choline PET/CT in comparison with CT and/or MRI in patients with hepatocellular carcinoma. Eur J Nucl Med Mol Imaging. 2015 Aug;42(9):1399-407. doi: 10.1007/s00259-015-3079-5. Epub 2015 May 12. PMID 25962590
- [Background] Talbot JN, Gutman F, Fartoux L, Grange JD, Ganne N, Kerrou K, Grahek D, Montravers F, Poupon R, Rosmorduc O. PET/CT in patients with hepatocellular carcinoma using [(18)F]fluorocholine: preliminary comparison with [(18)F]FDG PET/CT. Eur J Nucl Med Mol Imaging. 2006 Nov;33(11):1285-9. doi: 10.1007/s00259-006-0164-9. Epub 2006 Jun 27. PMID 16802155
- [Background] Lanza E, Donadon M, Felisaz P, Mimmo A, Chiti A, Torzilli G, Balzarini L, Lopci E. Refining the management of patients with hepatocellular carcinoma integrating 11C-choline PET/CT scan into the multidisciplinary team discussion. Nucl Med Commun. 2017 Oct;38(10):826-836. doi: 10.1097/MNM.0000000000000719. PMID 28723716
- [Background] Castello, A., Lopci, E. Imaging HCC treated with radioembolization: review of the literature and clinical examples of choline PET utility. Clin Transl Imaging (2020). https://doi.org/10.1007/s40336-020-00384-y